CLINICAL TRIAL: NCT06740916
Title: Long-term Efficacy of Once Daily Versus Twice Daily Aspirin in High-risk Myeloproliferative Neoplasms Patients with Aspirin Resistance
Brief Title: Long-term Efficacy of Once Daily Versus Twice Daily Aspirin in High-risk MPN Patients with Aspirin Resistance
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Yingyong Chinthammitr, Assistant Professor, Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Siriraj Hospital
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Myeloproliferative Neoplasms (MPN)
Keywords: myeloproliferative neoplasm; aspirin resistance
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 81-mg aspirin once daily (Active Comparator): 81-mg aspirin once daily
  Interventions: Drug: 81-mg aspirin once daily
- 81-mg aspirin twice daily (Experimental): 81-mg aspirin twice daily
  Interventions: Drug: 81-mg aspirin twice daily

INTERVENTIONS:
Drug: 81-mg aspirin once daily — 81-mg aspirin once daily
  Arms: 81-mg aspirin once daily
Drug: 81-mg aspirin twice daily — 81-mg aspirin twice daily
  Arms: 81-mg aspirin twice daily

SUMMARY:
Patients with myeloproliferative neoplasm (MPN) could have laboratory aspirin resistance and then increasing dose of aspirin from once daily to twice daily regimen is suggested. However, it is not routinely recommended to perform platelet function testing to determine aspirin resistance in MPN patients. Moreover, it is not known whether increasing dose of aspirin would always correct aspirin resistance and significantly prevent the thrombotic events in MPN patients. Therefore, this study aims to compare the efficacy of once daily versus twice daily aspirin in high-risk MPN patients with aspirin resistance. MPN patients with laboratory aspirin resistance will be included in this prospective randomized study and platelet function testing will be repeated at one and six months later. Clinical thrombosis and side effect from aspirin will be recorded for at least 2 years after intervention.

DETAILED DESCRIPTION:
Inclusion criteria included adult (>=18 years) Philadelphia-negative MPN patients taking aspirin (81 mg/day). Exclusion criteria included concomitant active cancer, thrombocytopenia (platelet less than 50,000/uL), taking anticoagulant, platelet function test (LTA method) showing no aspirin resistance, active gastric disease, active bleeding. Termination criteria included not taking aspirin regularly, serious side effect from aspirin. Block of four randomization is used. LTA testing is repeated at month 1 and 6 in both arms. PFA200 method is also done at initial enrollment for comparison with LTA method. Follow-up outcome data of clinical thrombosis, bleeding complication and adverse events related with aspirin are collected. Comparative analysis of outcome data is performed between two arms.

ELIGIBILITY:
Inclusion Criteria:

* Philadelphia negative Myeloproliferative neoplasms aged at least 18 years old

Exclusion Criteria:

* Concomitant other active malignancy or cured less than 6 months
* Platelet count less than 50,000/microL
* Receiving anticoagulant
* Active peptic ulcer
* Active bleeding or Planning to undergo procedure/operation with bleeding risk
* No laboratory aspirin resistance with LTA method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
prevalence of aspirin resistance | At 1 month and 6 month after intervention
  Laboratory aspirin resistance is determined by light transmission aggregometry using arachidonic acid (0.5 g/L) as agonist and result of aggregation >= 20% is defined as resistance.

SECONDARY OUTCOMES:
The incidence of thrombotic events | 2 years
  The thrombotic events will be recorded for at least 2 years after intervention.

OTHER OUTCOMES:
The cut-of-point of PFA200 to define aspirin resistance | At enrollment
  The standard definition of aspirin resistance in this study is determined by light transmission aggregometry (LTA) using arachidonic acid (0.5 g/L) as agonist and the result of aggregation of >=20% is defined as aspirin resistance. PFA200 is used in parallel with LTA method to determine the concordance of these two methods and to determine the appropriate cut-of-point of PFA200 method to define aspirin resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Hematology, Department of Medicine, Faculty of Medicine Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
basic characteristic
Supporting Information: Study Protocol, CSR
Time Frame: 1 Jan 2027 (start date) to 31 March 2027 (end date)
Access Criteria: Hematologists in academic centers, basic characteristic and result, contact via my email address

REFERENCES:
- [Background] Rocca B, Tosetto A, Petrucci G, Rossi E, Betti S, Soldati D, Iurlo A, Cattaneo D, Bucelli C, Dragani A, Di Ianni M, Ranalli P, Palandri F, Vianelli N, Beggiato E, Lanzarone G, Ruggeri M, Carli G, Elli EM, Renso R, Randi ML, Bertozzi I, Loscocco GG, Ricco A, Specchia G, Vannucchi AM, Rodeghiero F, De Stefano V, Patrono C; Aspirin Regimens in EsSential thrombocythemia (ARES) Investigators. Long-term pharmacodynamic and clinical effects of twice- versus once-daily low-dose aspirin in essential thrombocythemia: The ARES trial. Am J Hematol. 2024 Aug;99(8):1462-1474. doi: 10.1002/ajh.27418. Epub 2024 Jun 15. PMID 38877813
- [Background] Rocca B, Tosetto A, Betti S, Soldati D, Petrucci G, Rossi E, Timillero A, Cavalca V, Porro B, Iurlo A, Cattaneo D, Bucelli C, Dragani A, Di Ianni M, Ranalli P, Palandri F, Vianelli N, Beggiato E, Lanzarone G, Ruggeri M, Carli G, Elli EM, Carpenedo M, Randi ML, Bertozzi I, Paoli C, Specchia G, Ricco A, Vannucchi AM, Rodeghiero F, Patrono C, De Stefano V. A randomized double-blind trial of 3 aspirin regimens to optimize antiplatelet therapy in essential thrombocythemia. Blood. 2020 Jul 9;136(2):171-182. doi: 10.1182/blood.2019004596. PMID 32266380
- [Background] Tsantes AE, Mantzios G, Giannopoulou V, Tsirigotis P, Bonovas S, Rapti E, Mygiaki E, Kartasis Z, Sitaras NM, Dervenoulas J, Travlou A. Monitoring aspirin treatment in patients with thrombocytosis: comparison of the platelet function analyzer (PFA)-100 with optical aggregometry. Thromb Res. 2008;123(1):100-7. doi: 10.1016/j.thromres.2008.03.008. Epub 2008 Apr 21. PMID 18430462
- [Background] Pascale S, Petrucci G, Dragani A, Habib A, Zaccardi F, Pagliaccia F, Pocaterra D, Ragazzoni E, Rolandi G, Rocca B, Patrono C. Aspirin-insensitive thromboxane biosynthesis in essential thrombocythemia is explained by accelerated renewal of the drug target. Blood. 2012 Apr 12;119(15):3595-603. doi: 10.1182/blood-2011-06-359224. Epub 2012 Jan 10. PMID 22234683
- [Background] Dillinger JG, Sideris G, Henry P, Bal dit Sollier C, Ronez E, Drouet L. Twice daily aspirin to improve biological aspirin efficacy in patients with essential thrombocythemia. Thromb Res. 2012 Jan;129(1):91-4. doi: 10.1016/j.thromres.2011.09.017. Epub 2011 Oct 19. No abstract available. PMID 22014557